CLINICAL TRIAL: NCT03119714
Title: A Placebo-controlled, Cross-over, Study to Assess the Efficacy of the Oral Mast Cell Inhibitor Pemirolast in Allergen-induced Airway Obstruction and Inflammation in Subjects With Allergic Asthma
Brief Title: Pemirolast in Allergen Challenge (PEMAG)
Acronym: PEMAG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to results from other studies regarding efficacy of pemirolast
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Unit for Chemistry II, Department of Medical Biochemistry, Karolinska Institutet (Unknown); Occupational and Environmental Medicine, Sahlgrenska UH, Gothenburg (Unknown); Div Clinical Pharmacology, Karolinska University Hospital (Unknown); Dept. Respiratory Medicine, University of Amsterdam, Amsterdam (Unknown)
Responsible Party: Principal Investigator, Barbro Dahlen, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PEMAG-2016-v2.3
Record Dates: First submitted 2016-11-11; First posted 2017-04-19 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Allergic Asthma
Keywords: bronchoprovocation; early-late asthmatic reaction; mast cell stabilizer; mast cell mediators; sputum eosinophils
MeSH Terms: interventions — pemirolast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pemirolast (Active Comparator): Pemirolast 200mg bid 14-16 days
  Interventions: Drug: Pemirolast
- Placebo Oral Tablet (Placebo Comparator): Matching placebo bid 14-16 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Pemirolast — Treatment with pemirolast 200 mg bid for 14-16 days
  Other Names: CRD 007
  Arms: Pemirolast
Drug: Placebo Oral Tablet — Treatment with placebo bid for 14-16 days
  Arms: Placebo Oral Tablet

SUMMARY:
The purpose of this study is to establish the influence of the non-steroidal candidate-drug pemirolast on allergen-induced airway obstruction and inflammation in allergic subjects with asthma. Pemirolast is an orally available inhibitor of the release of mast cell mediators. The study will therefore test the hypothesis that global inhibition of the mast cell, resulting in decreased production of most of its mediator molecules, will provide a highly significant anti-asthmatic effect.

DETAILED DESCRIPTION:
This is a crossover randomized double blind, placebo-controlled study where the early and late response to allergen inhalation challenge will be compared during two treatment periods, with pemirolast 200 mg bid for 14 (to 16) days and matching placebo, respectively. Non-smoking female and male subjects (n = 12-15) with intermittent atopic asthma, requiring only β2-agonists to treat their asthma, will be recruited. A total of twelve subjects who demonstrate an early and a late asthmatic response to inhaled allergen challenge are required to complete the study for the primary end-point. The sample size is sufficient according to experience from a large number of studies and published power calculations of the model. The effects of pemirolast have never been studied before in an allergen provocation model. Primary variable is the effect of treatment on the mean maximum fall in forced expiratory volume in one second (FEV1) during the early and the late asthmatic reactions induced by allergen. Secondary variables are the effect on mast cell activation and airway inflammation measured as the urinary excretion of metabolites of prostaglandins and other lipid mediators and the percentage of sputum eosinophils, respectively. Tertiary variables are the effect of treatment on airway responsiveness expressed as the provocative dose of methacholine causing 20 per cent decrease in FEV1 (PD20FEV1), as well as biomarkers of airway inflammation in saliva, sputum, exhaled air and blood.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years inclusive
* Diagnosed asthma as defined by at least one of the following:

  * response to standard asthma treatment
  * episodic wheezing
  * change in lung function over short periods of time
* Non-smoker for the past two years and a total of smoking less than 5 pack-years
* Stable intermittent asthma, only using bronchodilator therapy as needed for the last 4 weeks
* FEV1 ≥ 75 % of predicted
* A positive skin prick test to pollen (grass, birch, mugwort) or animal dander (dog, cat) and a history of associated symptoms on exposure.

Exclusion Criteria:

* Any significant respiratory disease, other than asthma.
* Subjects with seasonal asthma may not be included if they are in their season and subjects allergic to animal dander must not have a pet on their own or similar close exposure.
* Use of:

  * Oral, injectable or inhaled glucocorticosteroid treatment for the last 4 weeks prior to inclusion or during the study
  * Inhaled long-acting β2-agonists, anticholinergic bronchodilators, antihistamines, theofyllines, nasal or inhaled cromones and antileukotrienes within 2 weeks of screening
  * Beta-blocking agents.
  * Immunomodulator drugs
  * NSAIDs.
* Upper or lower respiratory tract infection within 4 weeks of screening
* Females who are pregnant, intend to be or who are lactating. Female subjects of childbearing potential who are not willing to use adequate contraceptive methods (measures as required by local requirements or practice) during participation in the trial until at least three days after last intake of study treatments. Male subjects not surgically sterilized, who or whose partner is not using adequate contraceptive methods (measures as required by local requirements or practice) during participation in the trial until at least three days after last intake of study drug.
* Subjects with BMI >30.
* Evidence (from clinical laboratory tests, physical examination or medical history) of hepatic disease (other than Gilbert´s Syndrome)
* Evidence (from physical examination or medical history) of any diseases that affects gastrointestinal absorption.
* A diagnosis of brittle asthma (rapid fluctuations in disease severity).
* Participation in other study in the four weeks prior to screening.
* Evidence of drug or alcohol abuse.
* History of having taken barbiturates or other drugs affecting the liver drug-metabolising enzymes within one month of the start of the trial.
* Blood donor during the last four months prior to study start and throughout the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-11; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Bronchoconstriction measured as fall in FEV1 during the early (EAR) and late (LAR) asthmatic reaction induced by allergen | After treatment with pemirolast or matching placebo for 14-16 days

SECONDARY OUTCOMES:
Mast cell activation measured as urinary excretion of metabolites of lipid mediators (prostaglandins,isoprostanes,leukotrienes,tromboxanes) | After treatment with pemirolast or matching placebo for 14-16 days
  Urine samples will be analysed with mass spectrometry (UPLC-MS/MS) and data presented as ng.mmol creatinine-1 for all metabolites
Airway inflammation measured as the percentage of sputum eosinophils | After treatment with pemirolast or matching placebo for 14-16 days
  Induced sputum will be collected 7 hours after the last inhaled allergen dose and percentage of eosinophils will be measured

OTHER OUTCOMES:
Airway responsiveness expressed as methacholine PD20FEV1 | After treatment with pemirolast or matching placebo for 14-16 days
  Change in methacholine responsiveness after the allergen challenge will be compared during the two treatment periods
Measurement of inflammatory biomarkers in saliva | After treatment with pemirolast or matching placebo for 14-16 days
  Saliva is collected before and after challenges to monitor activation of mast cells and other inflammatory pathways
Measurement of biomarkers in blood | After treatment with pemirolast or matching placebo for 14-16 days
  Venous blood samples are collected at clinic visits for asthma biomarkers. Biomarkers are taken before and after challenges according to sub-protocols specific for each analyte.
Measurement of biomarkers in sputum | After treatment with pemirolast or matching placebo for 14-16 days
  Sputum induction is performed on particular study days to assess inflammatory cell content and to collect sputum supernatant for analysis of biomarkers.
Measurement of biomarkers in exhaled breath samples | After treatment with pemirolast or matching placebo for 14-16 days
  Collection of exhaled air using the eNose will be used for exploratory studies of specific volatile and particular components of the exhaled breath

CONTACTS AND LOCATIONS:
Overall Officials: Barbro Dahlén, MD,PhD, Principal Investigator — Lung and Allergy Clinic, Karolinska UH
Locations (1):
- Lung and Allergy Research Unit C2-88 Karolinska University Hospital Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Not planing to share data